CLINICAL TRIAL: NCT04600024
Title: The Importance of Pelvic Morphometric Measurements in Piriformis Syndrome: A Case-control Study
Brief Title: Pelvic and Hip Morphometry in Piriformis Syndrome
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FSMEAH
Record Dates: First submitted 2020-10-18; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Piriformis Muscle Syndrome; Anthropometry
Keywords: Anthropometry; Pelvic Bones; Muscle Syndrome, Piriformis; Prospective Studies; Case-Control Studies; femur neck / pathology
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Piriformis syndrome group: Patients who were diagnosed as PS by diagnostic injection with ultrasound guidance
  Interventions: Diagnostic Test: Ultrasound guided diagnostic injection
- Age and sex match control group: Patients who were excluded from the diagnosis of PS and had anteroposterior (AP) direct radiographic imaging

INTERVENTIONS:
Diagnostic Test: Ultrasound guided diagnostic injection — 4 cc lidocaine %2 injection into the piriformis muscle was performed for the diagnosis of piriformis syndrome. It was performed by the ultrasound-guidance to increase the accuracy of the injection.
  Groups: Piriformis syndrome group

SUMMARY:
In this case-control study, 23 patients diagnosed as PS by diagnostic injection with ultrasound guidance were selected as the study group. 22 patients who were excluded from the diagnosis of PS and had anteroposterior (AP) direct radiographic imaging were evaluated as the control group. On the AP Pelvic graph, the femoral neck-shaft angle, the distances between predetermined bony landmarks were measured blindly without knowing the diagnosis, and the findings were compared statistically.

This study aims to evaluate whether the anatomical structure of the pelvis predisposes to the etiopathogenesis of the piriformis syndrome.

DETAILED DESCRIPTION:
Piriformis syndrome (PS) is a neuromuscular disorder consisting of pain and symptoms caused by compression of the sciatic nerve and other structures that pass under the piriformis muscle (PM). Due to difficulties in diagnosis, PS is confused with other pathologies such as lumbar disc pathology, lumbosacral radiculopathy, and sacroiliac dysfunction. As a result, patients are exposed to unnecessary and ineffective treatments, even surgery. The main problems in the PS diagnosis are the absence of objective physical examination findings, radiological findings, and a clear etiology. When the pathophysiology and etiology of PS are considered, there is no identifiable cause in most patients. Previous studies suggest that trauma, anatomical variations, and the trigger point in the muscle may cause PS. No study in the literature radiologically examined the pelvis or hip bone morphological features in PS to the best of our knowledge. This study aims to determine whether pelvic or hip bone morphology features pose a risk for PS in this study.

ELIGIBILITY:
For Piriformis syndrome group (study group);

Inclusion Criteria:

* A dramatic relief of pain following piriformis muscle local anesthetic injection

Exclusion Criteria:

* Having a neurological deficiency
* Having lumbar, sacroiliac, hip, and thoracolumbar pathology (inflammatory or degenerative)
* Operation history at the lumbar and hip region
* Being in the gestational or lactational period
* Body mass index of greater than 35
* History of inflammatory or infectious disease
* Active psychiatric illness, severe systemic, vascular or malign disease

For the control group

Inclusion criteria:

-Having Anteroposterior pelvic radiographs for other medical reasons

Exclusion criteria:

* Having a present piriformis syndrome or a history of piriformis syndrome
* Having a neurological deficiency
* Having lumbar, sacroiliac, hip, and thoracolumbar pathology (inflammatory or degenerative)
* Operation history at the lumbar and hip region
* Being in the gestational or lactational period
* Body mass index of greater than 35
* History of inflammatory or infectious disease
* Active psychiatric illness, severe systemic, vascular or malign disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The physical medicine and rehabilitation outpatient clinic of Fatih Sultan Mehmet Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Femoral Neck-Shaft Angle (NSA) | The measurement was evaluated by two different investigators immediately after the pelvis anteroposterior radiography was taken.
  The NSA, also called caput collum-diaphyseal angle or inclination angle, defined as the angle between the longitudinal femoral shaft axis and femoral head-neck axis.
Posterior Superior Iliac Spine (PSIS)- Trochanter Major (TM) | The measurement was evaluated by two different investigators immediately after the pelvis anteroposterior radiography was taken.
  The distance between the posterior superior iliac spine and the greater trochanter
PSIS-Ischial Tuberosity (IT) | The measurement was evaluated by two different investigators immediately after the pelvis anteroposterior radiography was taken.
  The distance between the posterior superior iliac spine and the apex of the ischial tuberosity
IT-TM | The measurement was evaluated by two different investigators immediately after the pelvis anteroposterior radiography was taken.
  The distance between the apex of the ischial tuberosity and the greater trochanter
Sacrum-TM | The measurement was evaluated by two different investigators immediately after the pelvis anteroposterior radiography was taken.
  The distance between the sacrum and the greater trochanter

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Güleç, MD, Study Director — Fatih Sultan Mehmet Training and Research Hospital; Ilknur Aktas, MD, Study Director — Fatih Sultan Mehmet Training and Research Hospital; Feyza Unlu Ozkan, MD, Study Chair — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Research and Traning Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirschner JS, Foye PM, Cole JL. Piriformis syndrome, diagnosis and treatment. Muscle Nerve. 2009 Jul;40(1):10-8. doi: 10.1002/mus.21318. PMID 19466717
- [Background] Jankovic D, Peng P, van Zundert A. Brief review: piriformis syndrome: etiology, diagnosis, and management. Can J Anaesth. 2013 Oct;60(10):1003-12. doi: 10.1007/s12630-013-0009-5. Epub 2013 Jul 27. PMID 23893704
- [Background] Hopayian K, Song F, Riera R, Sambandan S. The clinical features of the piriformis syndrome: a systematic review. Eur Spine J. 2010 Dec;19(12):2095-109. doi: 10.1007/s00586-010-1504-9. Epub 2010 Jul 3. PMID 20596735
- [Background] Papadopoulos EC, Khan SN. Piriformis syndrome and low back pain: a new classification and review of the literature. Orthop Clin North Am. 2004 Jan;35(1):65-71. doi: 10.1016/S0030-5898(03)00105-6. PMID 15062719
- [Background] Probst D, Stout A, Hunt D. Piriformis Syndrome: A Narrative Review of the Anatomy, Diagnosis, and Treatment. PM R. 2019 Aug;11 Suppl 1:S54-S63. doi: 10.1002/pmrj.12189. Epub 2019 Jul 22. PMID 31102324
- [Background] Benson ER, Schutzer SF. Posttraumatic piriformis syndrome: diagnosis and results of operative treatment. J Bone Joint Surg Am. 1999 Jul;81(7):941-9. PMID 10428125
- [Background] Pace JB, Henning C. Episacroiliac lipoma. Am Fam Physician. 1972 Sep;6(3):70-3. No abstract available. PMID 4262540
- [Background] Coskun Benlidayi I, Guzel R, Basaran S, Aksungur EH, Seydaoglu G. Is coxa valga a predictor for the severity of knee osteoarthritis? A cross-sectional study. Surg Radiol Anat. 2015 May;37(4):369-76. doi: 10.1007/s00276-014-1359-6. Epub 2014 Aug 12. PMID 25113012
- [Result] Durrani Z, Winnie AP. Piriformis muscle syndrome: an underdiagnosed cause of sciatica. J Pain Symptom Manage. 1991 Aug;6(6):374-9. doi: 10.1016/0885-3924(91)90029-4. PMID 1880438
- [Result] Hopayian K, Danielyan A. Four symptoms define the piriformis syndrome: an updated systematic review of its clinical features. Eur J Orthop Surg Traumatol. 2018 Feb;28(2):155-164. doi: 10.1007/s00590-017-2031-8. Epub 2017 Aug 23. PMID 28836092
- [Result] Kean Chen C, Nizar AJ. Prevalence of piriformis syndrome in chronic low back pain patients. A clinical diagnosis with modified FAIR test. Pain Pract. 2013 Apr;13(4):276-81. doi: 10.1111/j.1533-2500.2012.00585.x. Epub 2012 Aug 2. PMID 22863240
- [Result] Hallin RP. Sciatic pain and the piriformis muscle. Postgrad Med. 1983 Aug;74(2):69-72. doi: 10.1080/00325481.1983.11698378. No abstract available. PMID 6878094
- [Result] Niu CC, Lai PL, Fu TS, Chen LH, Chen WJ. Ruling out piriformis syndrome before diagnosing lumbar radiculopathy. Chang Gung Med J. 2009 Mar-Apr;32(2):182-7. PMID 19403008
- [Result] Rodrigue T, Hardy RW. Diagnosis and treatment of piriformis syndrome. Neurosurg Clin N Am. 2001 Apr;12(2):311-9. PMID 11525209
- [Result] Misirlioglu TO, Akgun K, Palamar D, Erden MG, Erbilir T. Piriformis syndrome: comparison of the effectiveness of local anesthetic and corticosteroid injections: a double-blinded, randomized controlled study. Pain Physician. 2015 Mar-Apr;18(2):163-71. PMID 25794202
- [Result] Haladaj R, Pingot M, Polguj M, Wysiadecki G, Topol M. Anthropometric Study of the Piriformis Muscle and Sciatic Nerve: A Morphological Analysis in a Polish Population. Med Sci Monit. 2015 Dec 2;21:3760-8. doi: 10.12659/msm.894353. PMID 26629744
- [Result] Guvencer M, Akyer P, Iyem C, Tetik S, Naderi S. Anatomic considerations and the relationship between the piriformis muscle and the sciatic nerve. Surg Radiol Anat. 2008 Aug;30(6):467-74. doi: 10.1007/s00276-008-0350-5. Epub 2008 May 6. PMID 18458807
- [Result] Menge TJ, Truex NW. Femoroacetabular impingement: a common cause of hip pain. Phys Sportsmed. 2018 May;46(2):139-144. doi: 10.1080/00913847.2018.1436844. Epub 2018 Feb 13. PMID 29406812
- [Result] Krueger DR, Windler M, Gesslein M, Schuetz M, Perka C, Schroeder JH. Is the evaluation of the anterior inferior iliac spine (AIIS) in the AP pelvis possible? Analysis of conventional X-rays and 3D-CT reconstructions. Arch Orthop Trauma Surg. 2017 Jul;137(7):975-980. doi: 10.1007/s00402-017-2694-y. Epub 2017 Apr 21. PMID 28432458
- [Result] Bredella MA, Azevedo DC, Oliveira AL, Simeone FJ, Chang CY, Stubbs AJ, Torriani M. Pelvic morphology in ischiofemoral impingement. Skeletal Radiol. 2015 Feb;44(2):249-53. doi: 10.1007/s00256-014-2041-0. Epub 2014 Nov 6. PMID 25371087
- [Result] Gomez-Hoyos J, Schroder R, Reddy M, Palmer IJ, Martin HD. Femoral Neck Anteversion and Lesser Trochanteric Retroversion in Patients With Ischiofemoral Impingement: A Case-Control Magnetic Resonance Imaging Study. Arthroscopy. 2016 Jan;32(1):13-8. doi: 10.1016/j.arthro.2015.06.034. Epub 2015 Sep 7. PMID 26358634
- [Result] Boese CK, Frink M, Jostmeier J, Haneder S, Dargel J, Eysel P, Lechler P. The Modified Femoral Neck-Shaft Angle: Age- and Sex-Dependent Reference Values and Reliability Analysis. Biomed Res Int. 2016;2016:8645027. doi: 10.1155/2016/8645027. Epub 2016 Dec 14. PMID 28070521
- [Result] Elbuken F, Baykara M, Ozturk C. Standardisation of the neck-shaft angle and measurement of age-, gender- and BMI-related changes in the femoral neck using DXA. Singapore Med J. 2012 Sep;53(9):587-90. PMID 23023899
- [Result] Gilligan I, Chandraphak S, Mahakkanukrauh P. Femoral neck-shaft angle in humans: variation relating to climate, clothing, lifestyle, sex, age and side. J Anat. 2013 Aug;223(2):133-51. doi: 10.1111/joa.12073. Epub 2013 Jun 19. PMID 23781912
- [Result] Fischer CS, Kuhn JP, Volzke H, Ittermann T, Gumbel D, Kasch R, Haralambiev L, Laqua R, Hinz P, Lange J. The neck-shaft angle: an update on reference values and associated factors. Acta Orthop. 2020 Feb;91(1):53-57. doi: 10.1080/17453674.2019.1690873. Epub 2019 Nov 18. PMID 31735107
- [Result] Fearon A, Stephens S, Cook J, Smith P, Neeman T, Cormick W, Scarvell J. The relationship of femoral neck shaft angle and adiposity to greater trochanteric pain syndrome in women. A case control morphology and anthropometric study. Br J Sports Med. 2012 Sep;46(12):888-92. doi: 10.1136/bjsports-2011-090744. Epub 2012 Apr 30. PMID 22547561